CLINICAL TRIAL: NCT04109586
Title: Preventing Neurogenic Obesity Following Traumatic Spinal Cord Injury
Brief Title: Diet and Fat Mass After Traumatic Spinal Cord Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: University of Oslo (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Vegard Strøm, Head of Research Group, Sunnaas Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REK 2017/2443
Record Dates: First submitted 2019-07-03; First posted 2019-09-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Metabolic Disease; Spinal Cord Injuries
MeSH Terms: conditions — Obesity; Metabolic Diseases; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized nutrition therapy (Experimental): Dietitian led assessment and individual nutritional therapy during inpatient rehabilitation with follow-up the first year after injury
  Interventions: Behavioral: Personalized nutritional therapy
- Standard treatment (No Intervention): Standard treatment includes dietitian-led group session on nutrition after SCI and patient visits / consultations on request from doctor.

INTERVENTIONS:
Behavioral: Personalized nutritional therapy — Dietitian led assessment and individual nutritional therapy during inpatient rehabilitation with follow-up the first year after injury
  Arms: Personalized nutrition therapy

SUMMARY:
This is a randomized clinical controlled trial (RCT) to investigate the impact of a personalized nutritional intervention on functional and clinical outcomes the first year after traumatic spinal cord injury. The long term goal is to prevent gain of body fat mass and obesity.

DETAILED DESCRIPTION:
Traumatic spinal cord injury (SCI) is a devastating injury resulting from critical incidents like falls, sports- and traffic accidents, demanding lifelong specialist health care services. A major challenge is the prevalence of obesity following metabolic alterations after SCI. Obesity hampers independence and mobility and has a negative impact on quality of life. Accumulation of adipose tissue is reported to be higher than in able-bodied, explaining the high risk of cardiometabolic disease in the SCI population. Food intake is the supreme variable in prevention of obesity after SCI, however there is a paucity in studies investigating nutrition as a measure to prevent and reduce comorbidity. Key questions that remains unanswered are how early adipose tissue accumulates, if nutritional manipulations can prevent obesity and how follow-up can help maintain a healthy lifestyle. In the present PhD-study, we use MRI techniques to quantify changes in body composition in a cohort study the first year after SCI, and we employ a randomized controlled trial to test the efficacy of a nutrition intervention during rehabilitation aiming to prevent obesity. Successful results will be implemented in care-programs at our hospital for those with SCI and similar mobility impairments, with the aim of improving nutrition practice throughout the course of treatment

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury
* Levels C1-L2
* American Spinal Injury Association (ASIA) Impairments Scale (AIS) A-D

Exclusion Criteria:

* Glasgow Coma Scale score (GCS) equal to or lower than 13
* Below 18 years of age
* Medical issues like impaired cognitive function, progressive disorders and co-morbidities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in fat mass (kg) | Change from Baseline to 12 months follow-up
  Bioimpedance analysis (BIA; seca mBCA 525) will be used to assess whole-body composition. Total fat mass (kg) derived from BIA will be used as the primary adiposity outcome. In individuals with spinal cord injury, fluid shifts and changes in fat-free mass can influence BIA estimates; therefore, fat mass will be interpreted together with secondary indices (fat mass index and waist circumference) and body water compartments.

SECONDARY OUTCOMES:
Change in Fat Mass Index (FMI, kg/m2) | Change from baseline to 12 months follow-up
  Fat mass index (FMI) will be calculated as total fat mass (kg) divided by height squared (m²), based on BIA-derived fat mass. FMI will be analysed as a key secondary adiposity index, as it standardizes fat mass for body size and may provide a more stable estimate of adiposity than absolute fat mass in spinal cord injury.
Change in BIA-estimated visceral adipose tissue | Change from baseline to 12 months follow-up
  Visceral adipose tissue (VAT) will be estimated using the manufacturer's proprietary prediction equations implemented in the seca mBCA 525. These values represent model-based estimates calibrated against MRI in able-bodied populations and are interpreted as surrogate indicators of central adiposity rather than direct imaging measures. VAT will be analysed as a secondary adiposity outcome.
Waist circumference (WC, cm) | Change from baseline to 12 months follow-up
  Waist circumference will be measured at the midpoint between the lower rib margin and the iliac crest (approximately 2 cm above the umbilicus) using a standardized protocol. Waist circumference is included as an anthropometric marker of central adiposity.
Change in Fat-free mass | Change from baseline to 12 months follow-up
  Fat-free mass (FFM) derived from BIA will be used to describe changes in lean tissue. In this population, FFM is strongly influenced by extracellular water shifts and will therefore be used as supportive information for interpreting changes in fat mass.
Body weight | Change from Baseline to 12 months follow-up
  Measuring body weight in kilograms (kg)
Body mass index (BMI, kg/m²) | Change from baseline to 12 months follow-up.
  Body mass index (kg/m²) will be calculated from weight and height according to standard procedures. BMI is included as an anthropometric indicator of overall adiposity.
Change in adipose tissue | Change from Baseline to 12 months follow-up
  Magnetic resonance imaging (MRI) scanning will be used to determine body composition by quantification of adipose tissues (visceral adipose tissue volume and abdominal subcutaneous adipose tissue volume) and muscle volumes.
Change in fasting blood glucose level (mmol/Liter) | Change from Baseline to 12 months follow-up
  Standardized oral glucose tolerance test (OGTT) will be used to measure the blood glucose level (mmol/Liter) 2 hours after intake of 75 grams glucose in a fasted state.
Change in fasting glucose | Change from Baseline to 12 months follow-up
  Fasted blood analysis of fasting glucose (mmol/L)
Change in Glycated hemoglobin (HbA1c) | Change from Baseline to 12 months follow-up
  Fasted blood analysis of HbA1c mmol/mol
Change in Cholesterol | Change from Baseline to 12 months follow-up
  Fasted blood analysis of total cholesterol, high density lipoprotein (HDL) and low density lipoprotein (LDL) mmol/L
Change in Triglycerides | Change from Baseline to 12 months follow-up
  Fasted blood analysis of triglycerides mmol/L
Changes in Quality of life (QoL) | Changes from Baseline to 12 months follow-up
  International Spinal Cord Society QoL Basic Dataset. The QoL data set consists of 3 variables: ratings of satisfaction with general quality of life, satisfaction with physical health, and satisfaction with psychological health. All variables are rated on a Numeric Self-Rating Scale ranging from 0 (completely dissatisfied) to 10 (completely satisfied).
Independency in activities of daily living (ADLs) | Change from Baseline to 12 months follow-up
  Spinal Cord Independence Measure (SCIM) III will be used to assess various activities of daily living (ADLs). SCIM III comprises 19 items divided into 3 subscales (self-care, respiration and sphincter management, and mobility). The total SCIM score range from 0 to 100, with the subscales weighted as follows: self-care: scored 0-20; respiration and sphincter management: scored 0-40; and mobility: scored 0-40. Scores are higher in patients that require less assistance or fewer aids to complete basic ADLs.
Change in albumin | Change from Baseline to 12 months follow-up
  Fasted blood analysis of albumin g/dl
Change in Creatinine | Change from Baseline to 12 months follow-up
  Fasted blood analysis of creatinine umol/L
Change in Lipoprotein A1 | Change from Baseline to 12 months follow-up
  Fasted blood analysis of Lipoprotein A1 (g/L)
Change in Lipoprotein B | Change from Baseline to 12 months follow-up
  Fasted blood analysis of Lipoprotein B (g/L)
Change in folic acid | Change from Baseline to 12 months follow-up
  Fasted blood analysis of folic acid (nmol/L)
Change in vitamin B12 | Change from Baseline to 12 months follow-up
  Fasted blood analysis of vitamin B12 pmol/L
Change in Ferritin | Change from Baseline to 12 months follow-up
  Fasted blood analysis of ferritin ug/L
Change in C-reactive protein (CRP) | Change from Baseline to 12 months follow-up
  Fasted blood analysis of C-reactive protein mg/l
Change in C-peptid | Change from Baseline to 12 months follow-up
  Blood analysis of insulin c-peptid pmol/L in a fasted state and 2 hours post oral glucose tolerance test
Change in vitamin 25-hydroxy-vitamin D₃ | Change from Baseline to 12 months follow-up
  Fasted blood analysis of 25-hydroxy-vitamin D₃ (nmol/L)
Change in Cytokines: Interleukin-6 and -1, Tumor necrosis factor-α (TNF-α) | Change from Baseline to 12 months follow-up
  Fasted blood analysis of Interleukin-6 and -1 Tumor necrosis factor-α (TNF-α) (pg/ml)
Change in isoprostanes (biomarkers of oxidative stress) | Change from Baseline to 12 months follow-up
  Urine analyses of isoprostanes (ng/mg) (biomarkers of oxidative stress)
Change in cardiorespiratory fitness levels ml/kg/min | Change from Baseline to 12 months follow-up
  Cardiorespiratory fitness levels will be determined by measuring peak oxygen uptake (VO2peak; ml/kg/min) during maximal exercise testing on a treadmill or ergometry cycle.
Change in cardiorespiratory fitness levels liter/min | Change from Baseline to 12 months follow-up
  Cardiorespiratory fitness levels will be determined by measuring peak oxygen uptake (VO2peak; liter/min) during maximal exercise testing on a treadmill or ergometry cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Strøm, PhD, Principal Investigator — Sunnaas Rehabilitation Hospital
Locations (1):
- Sunnaas Rehabilitation Hospital, Nesoddtangen, Bjørnemyr, Norway

IPD SHARING:
Plan to Share IPD: No